CLINICAL TRIAL: NCT05423717
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Polysomnography, Dose-finding Study Assessing the Efficacy, Safety, and Pharmacokinetics of Multiple-dose Oral Administration of Daridorexant in Pediatric Subjects Aged 10 to < 18 Years With Insomnia Disorder
Brief Title: Dose-finding Study Assessing the Efficacy, Safety, and Pharmacokinetics of Daridorexant in Subjects Aged 10 to < 18 Years With Insomnia Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-078A205; 2024-513885-20-00 (EU CTIS Number)
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-05

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Daridorexant 10 mg (Experimental)
  Interventions: Drug: Daridorexant 10 mg
- Daridorexant 25 mg (Experimental)
  Interventions: Drug: Daridorexant 25 mg
- Daridorexant 50 mg (Experimental)
  Interventions: Drug: Daridorexant 50 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daridorexant 10 mg — Daridorexant will be taken orally, once daily in the evening during the treatment period.
  Arms: Daridorexant 10 mg
Drug: Daridorexant 25 mg — Daridorexant will be taken orally, once daily in the evening during the treatment period.
  Arms: Daridorexant 25 mg
Drug: Daridorexant 50 mg — Daridorexant will be taken orally, once daily in the evening during the treatment period.
  Arms: Daridorexant 50 mg
Drug: Placebo — Placebo will be taken orally, once daily in the evening during the treatment period.
  Arms: Placebo

SUMMARY:
This study assesses the efficacy, safety, and pharmacokinetics of multiple-dose oral administration of daridorexant in pediatric subjects aged 10 to < 18 years with insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form (ICF) from the caregiver, i.e., parent/legal guardian prior to any study mandated procedure, or as per local regulation.
* Written assent must be obtained from subjects of the appropriate age who can give assent, as determined by the caregiver and local regulation or institutional review boards / independent ethics committees.
* Male or female subjects aged ≥ 10 and < 18 years at the time of signing the ICF.
* Chronic insomnia disorder in accordance with International Classification of Sleep Disorders, 3rd edition (ICSD-3) or insomnia disorder in accordance with Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria at Screening, as supported by statements from the child and/or the caregiver:

  1. Difficulty initiating or maintaining sleep, or early morning awakening with inability to return to sleep,
  2. Sleep difficulty has been present for at least 3 months prior to Screening,
  3. Sleep difficulty occurs at least 3 nights per week,
  4. Persistence of sleep difficulty, despite adequate sleep hygiene or non-pharmacological therapy,
  5. The sleep problem occurs despite adequate age appropriate time and opportunity for sleep,
  6. The sleep problem is not due to the direct pharmacological effects of any concomitant medication (e.g., amphetamines, selective serotonin reuptake inhibitors) as per investigator judgment,
  7. Self-report or caregiver report of poor sleep quality and/or quantity impacting the daytime performance of the subject,
* Sleep Disturbance Scale for Children score > 16 on the Difficulty Initiating or Maintaining Sleep domain at Screening.
* Adolescent of Child-Bearing Potential:

  1. Negative serum pregnancy test at Screening and a negative urine pregnancy test at Randomization.
  2. Agreement to undertake urine pregnancy tests during the study, as per the schedule of activities and up to 5 days after study treatment discontinuation.
  3. Agreement to use an acceptable effective method of contraception from Screening up to 5 days after study treatment discontinuation.
* Inclusion criteria applicable only to a subset of children with insomnia and comorbid neurodevelopmental disorder (NDD): Must have a documented history of NDD (including autism spectrum disorder or attention deficit hyperactivity disorder) according to DSM-5 criteria, as confirmed by review of medical records, at Screening. Use of central nervous system (CNS) stimulants is allowed if started at least 4 weeks prior to Screening, is stable, and is expected to remain stable during the study until End-of-Treatment. CNS stimulants are recommended to be taken in the morning.

Exclusion Criteria:

* Body weight < 25 kg.
* Daytime napping ≥ 1 h per day on at least 3 weekdays per week during the 3 months prior to Screening.
* Any lifetime history of sleep-related breathing disorders such as obstructive sleep apnea, based on the subject's medical records. Note: a subject whose breathing disorder has been treated by tonsillectomy/ adenoidectomy remains eligible.
* Any other diagnosed sleep-wake disorder as defined in DSM-5 or ICSD-3 (e.g., restless legs syndrome, circadian rhythm sleep wake disorder, parasomnias, narcolepsy) at Screening.
* Any of the following conditions related to suicidality:

  1. Any suicidal ideation with intent, with or without a plan at Screening, i.e., answering "Yes" to questions 4 or 5 on the suicidal ideation section of the lifetime (Visit 1) and visit (Visit 2) version of the Columbia Suicide Severity Rating Scale© (C-SSRS©). Participants who answer "yes" to any of these questions must be referred to the investigator for follow-up evaluation.
  2. History of suicide attempt on the suicidal behavior section of the lifetime version of the C-SSRS© at Visit 1.
* Any acute or unstable significant medical condition (e.g., seizure disorder, bipolar disorder, schizophrenia), hematology/biochemistry test results, and/or electrocardiogram results deviating from the normal ranges to a clinically relevant extent that would preclude participation in the study or could prevent the subject from complying with study requirements, as per investigator judgement.
* Cognitive behavior therapy for any indication is allowed only if it has been started at least 1 month prior to Visit 2 and is kept stable throughout the study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Day 1 in Total Sleep Time (TST) as measured by polysomnography (PSG). | PSG will be performed on 2 nights during the screening period and on Day 1 of the treatment period (total duration: 3 days).
  Baseline is defined as the mean of the 2 PSG nights during the screening period.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (35):
- United States (12):
  - Banner - University Medical Center Tucson, Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Teradan Clinical Trials, Brandon, Florida
  - D&H National Research Centers, Inc., Miami, Florida
  - Hope Research Network, Miami, Florida
  - University of South Florida - Tampa General Hospital (TGH), Tampa, Florida
  - Encore Medical Research of Weston, Weston, Florida
  - Florida Pediatric Research Institute, Winter Park, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - National Clinical Research, Inc, Richmond, Virginia
- Bulgaria (8):
  - MC Zdrave 1 Ltd., Kozloduy
  - MHAT "Heart and Brain" (SJSC), Pleven
  - University Hospital (UMHAT) Sveti Georgi, Plovdiv
  - MC ReSpiro Ltd., Razgrad
  - MC Sun I Zdrave ("Sleep and health") Ltd., Sofia
  - MC Kalimat, Sofia
  - MC Inspiro, Sofia
  - MC Sanamedik Ltd., Varna
- Germany (5):
  - Advanced Sleep Research Berlin GmbH, Berlin
  - Charité -Universitätsmedizin Berlin, Berlin
  - Vestische Caritas-Kliniken GmbH, Vestische Kinder- und Jugendklinik Datteln, Datteln
  - ProSomno, München
  - SOMNIBENE Institut für Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin
- Italy (3):
  - IRCCS Ospedale Bellaria, Bologna
  - Meyer Children's Hospital, Florence
  - Institute Giannina Gaslini, Genova
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - HM Puerta del Sur, Unidad del Sueño, Móstoles
  - Hospital Quironsalud Valencia - Sleep Unit, Valencia
  - Hospital Universitario Araba, Vitoria-Gasteiz
- Switzerland (2):
  - Universitäts-Kinderspital beider Basel (UKBB), Basel
  - Ospedale Regionale di Lugano Civico - Neurocentro della Svizzera Italiana, Sleep Medicine Unit, Lugano

IPD SHARING:
Plan to Share IPD: No